CLINICAL TRIAL: NCT04297631
Title: Prospective Study Investigating Antibiotic Elution From Free Intra-articular Vancomycin and Tobramycin After Cementless Total Knee Arthroplasty
Brief Title: Intraarticular Antibiotic in TKA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201911147
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Results first posted 2021-10-05 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Antibotics in Cementless Knees

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Vancomycin Powder (Experimental): All patients getting vancomycin to see concentration after 24hrs in knee drain and serum levels.
  Interventions: Device: Vancomyscin
- Tobramycin Powder (Experimental): All patients getting Tobramycin to see conceration after 24hrs in knee drain and serum levels.
  Interventions: Drug: Tobramycin Powder

INTERVENTIONS:
Drug: Tobramycin Powder — Everyone gets tobramycin powder.
  Arms: Tobramycin Powder
Device: Vancomyscin — Everyone gets the vancomyscin powder.
  Arms: Vancomycin Powder

SUMMARY:
The purpose of the study is to determine the intra-articular concentration of vancomycin and tobramycin after administration of vancomycin and tobramycin powder in primary cementless total knee arthroplasty and determine the serum concentrations of these antibiotics postoperatively.

DETAILED DESCRIPTION:
Patients will be identified by medical record review to make sure they meet inclusion and exclusion criteria. Patients that qualify and sign consent will have tobramycin and vancomycin antibiotic powder placed into the knee during surgery. Postoperative drain fluid from the knee will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18
2. Total knee arthroplasty for primary osteoarthritis. Primary diagnosis of knee osteoarthritis

Exclusion Criteria:

1. Diminished mental capacity
2. Vancomycin allergy
3. Tobramycin allergy
4. Chronic kidney disease stage III and stage IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-11-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Vancomycin: All patients getting vancomycin and tobramycin to see concentration after 24hrs in knee drain and serum levels.
  Vancomyscin: Everyone gets the vancomyscin powder.
  Tobramycin Powder: Everyone gets tobramycin powder.
Period: Overall Study
Arm/Group | Vancomycin
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Vancomycin
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Vancomycin [Count of Participants; unit: Participants] — All patients getting vancomycin and tobramycin to see concentration after 24hrs in knee drain and serum levels.
  Vancomyscin: Everyone gets the vancomyscin powder. Tobramycin Powder: Everyone gets tobramycin powder.
  Participants | 20

OUTCOME MEASURES:

1. Primary Outcome: Concentration of Antibiotics in Cementless Knees Post op
Description: 1. Determine the intra-articular concentration of vancomycin and tobramycin after administration of vancomycin and tobramycin powder in primary cementless total knee arthroplasty.
Time Frame: 1 hour, 4 hours, and 24 hours
Population: All primary cementless TKA two surgeons at a single institution over a 4-week period were assessed preoperatively for study inclusion.
Measure: Median (Full Range); unit: micrograms per milliliter
Groups:
- Intraarticular Concentrations of Tobramycin and Vancomycin: All patients getting vancomycin and tobramycin to see serum concentration after 24hrs in knee drain and serum levels.
  Vancomyscin: Everyone gets the vancomyscin powder.
  Tobramycin Powder: Everyone gets tobramycin powder.
Arm/Group | Intraarticular Concentrations of Tobramycin and Vancomycin
Number analyzed (Participants) | 20
micrograms per milliliter
  1 hour Vancomycin Intraarticular concentration | 1702.5 [440 to 4000]
  4 hour Vancomycin Intraarticular concentration | 582.5 [61 to 2400]
  24 hour Vancomycin Intraarticular concentration | 56.1 [12.4 to 290]
  1 hour tobramycin Intraarticular concentration | 1943 [345 to 7850]
  4 hour tobramycin Intraarticular concentration | 345 [31.8 to 1150]
  24 hour tobramycin Intraarticular concentration | 8.7 [1.5 to 358]

2. Secondary Outcome: Serum Concentrations of Vancomycin and Tobramycin at 1, 4, and 24 Hours.
Description: 2. Determine the serum concentrations of these antibiotics postoperatively
Time Frame: 1 hour, 4 hours, and 24 hours
Measure: Median (Full Range); unit: micrograms per milliliter
Groups:
- Vancomycin and Tobramycin Serum Concentration: All patients getting vancomycin and tobramycin to see concentration after 24hrs in knee drain and serum levels.
  Vancomyscin: Everyone gets the vancomyscin powder.
  Tobramycin Powder: Everyone gets tobramycin powder.
Arm/Group | Vancomycin and Tobramycin Serum Concentration
Number analyzed (Participants) | 20
micrograms per milliliter
  1 hour vancomycin serum concentration | 2.3 [0 to 3.9]
  4 hour vancomycin serum concentration | 4.6 [0 to 6.8]
  24 hour vancomycin serum concentration | 3.1 [0 to 5.8]
  1 hour tobramycin serum concentration | 6.3 [3.2 to 8.4]
  4 tobramycin | 8 [3.1 to 10.5]
  24 hour tobramycin | .8 [0.5 to 2]

ADVERSE EVENTS:
Time Frame: Adverse events were captured while patient was in hospital which was about 24 hours.
Description: study involved collecting fluid and blood from patients at post-op timepoints.
Arm/Group | Intraarticular Concentrations of Tobramycin and Vancomycin
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-10): https://cdn.clinicaltrials.gov/large-docs/31/NCT04297631/Prot_SAP_000.pdf
  • Informed Consent Form (2020-02-13): https://cdn.clinicaltrials.gov/large-docs/31/NCT04297631/ICF_001.pdf